CLINICAL TRIAL: NCT03087370
Title: A Retrospective and Prospective Natural History Study of Patients With WHIM Syndrome
Status: Withdrawn | Type: Observational
Why Stopped: Company Decision
Sponsor: X4 Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: X4-WHIM-NTHX
Record Dates: First submitted 2017-03-10; First posted 2017-03-22 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: WHIM Syndrome
Keywords: CXCR4 Mutation; Primary immunodeficiency disorder; Warts; Hypogammaglobulinemia; Infections; Myelokathexis; Human papillomavirus (HPV); Neutropenia; Herpes
MeSH Terms: conditions — WHIM syndrome; Primary Immunodeficiency Diseases; Warts; Agammaglobulinemia; Infections; Neutropenia; Herpes Simplex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood or buccal swab for the purposes of identifying a CXCR4 mutation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This natural history study is a prospective and retrospective, observational study of WHIM patients. WHIM syndrome is a rare, genetic, primary immunodeficiency disorder (a disorder in which the body's immune system does not function properly). WHIM is an acronym for some of the symptoms of the disorder - Warts, Hypogammaglobulinemia (low levels of certain antibodies), Infections and Myelokathexis (too many white blood cells in the bone marrow).This study includes 10-year retrospective (Retrospective Phase) and up to 5-year prospective (Prospective Phase) components.

DETAILED DESCRIPTION:
Given the rarity of patients with WHIM syndrome, this study is being conducted to better understand the clinical course of untreated patients with WHIM syndrome.

The goals of this Natural History Study are to define both the frequency and diversity of WHIM syndrome by specific genetic mutation, as well as to understand the clinical course and phenotype of untreated WHIM patients.

ELIGIBILITY:
Inclusion Criteria:

1. Has a confirmed clinical diagnosis of WHIM syndrome.
2. Has signed the current approved informed consent form; patients under 18 years of age will sign an approved informed assent form and must also have a signed parental consent.
3. Be willing and able to comply with the study protocol.

Exclusion Criteria:

1. Has, within 6 months prior to Day 1, received a CXCR4 antagonist.
2. Currently participating in an investigational study for treatment of WHIM.
3. Has any other medical or personal condition that, in the opinion of the Investigator, may potentially compromise the safety or compliance of the patient, or may preclude the patient's successful completion of the clinical study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnoses with WHIM syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of infections | Up to five years, from time of enrollment through study completion or early termination
  Infections assessed by hospitalizations (including intensive care), antibiotic use, outpatient medical appointments and missed days of school/work.
Severity of infections | Up to five years, from time of enrollment through study completion or early termination
Incidence of warts | Up to five years, from time of enrollment through study completion or early termination
Severity of warts | Up to five years, from time of enrollment through study completion or early termination
  Warts assessed by number and size of lesions, need for surgical, systemic or topical treatment and complications.
Change in quality of life over time | Up to five years, from time of enrollment through study completion or early termination
  Quality of life as assessed by the quality of life instrument the 36-Item Short Form Survey (SF-36)
Change in quality of life over time | Up to five years, from time of enrollment through study completion or early termination
  Quality of life as assessed by the quality of life instrument the Pediatric Quality of Life Inventory (Peds-QL)
Change in quality of life over time | Up to five years, from time of enrollment through study completion or early termination
  Quality of life as assessed by the quality of life instrument the Life Quality Index (LQI)
Change in quality of life over time | Up to five years, from time of enrollment through study completion or early termination
  Quality of life as assessed by the quality of life instrument the HPV Impact Profile (HIP)
Change in medical resource utilization | Up to five years, from time of enrollment through study completion or early termination
Change in absolute neutrophil count (ANC) over time | Up to five years, from time of enrollment through study completion or early termination
Change in absolute lymphocyte count (ALC) over time | Up to five years, from time of enrollment through study completion or early termination
Change in serum immunoglobulin over time | Up to five years, from time of enrollment through study completion or early termination
Changes in anti-vaccine antibodies over time | Up to five years, from time of enrollment through study completion or early termination

CONTACTS AND LOCATIONS:
Overall Officials: Sudha Parasuraman, MD, Study Director — X4 Pharmaceuticals, Inc.

IPD SHARING:
Plan to Share IPD: Yes